CLINICAL TRIAL: NCT06881199
Title: Complete Denture Palatal Material Impact on Patients' Satisfaction and Oral Health-Related Quality of Life: a Randomized Crossover Clinical Trial
Brief Title: "Acrylic Vs. Metal Palatal Coverage in Complete Dentures: Patient-Reported Outcomes"
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Motasum Abu-Awwad, Associate Professor, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 10/2024/10664
Record Dates: First submitted 2024-05-03; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Complete Edentulism; Satisfaction, Patient; Quality of Life
MeSH Terms: conditions — Patient Satisfaction | interventions — Denture, Complete

STUDY DESIGN:
Intervention Model Description: Patients will randomly be allocated to either group A/B or B/A. Group A: Patients receiving an acrylic complete denture Group B: Patients receiving a metal palate complete denture
  After insertion, all participants will be followed up for a minimum of 1 week to correct any issues with the dentures and eliminate patient complaints.
  All patients will be recalled at 2 month after insertion to answer questions using the VAS and to fill out the Oral Health Impact Profile-20 EDENT (OHIP-EDENT), and receive the other type of palatal material.
  After the second period the same process will be repeated.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not be aware of which group he/she is interviewing at the assessment session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acrylic palate complete denture (Experimental): Participants will receive maxillary complete dentures with an acrylic palate
  Interventions: Other: Complete denture with a metallic Co-Cr casted palate
- Metal palate complete denture (Experimental): Participants will receive maxillary complete dentures with a metal palate
  Interventions: Other: Complete denture with an acrylic palate

INTERVENTIONS:
Other: Complete denture with a metallic Co-Cr casted palate — Complete denture with a metallic Co-Cr casted palatal material
  Other Names: Complete denture with an acrylic palate
  Arms: Acrylic palate complete denture
Other: Complete denture with an acrylic palate — Complete denture with an acrylic palatal material
  Arms: Metal palate complete denture

SUMMARY:
Conventional dentures can be uncomfortable and limit oral functionality due to the polished surfaces covering the palate and rugae areas. A randomized crossover clinical trial was conducted to compare patients' satisfaction and oral health-related quality of life when using dentures with an acrylic or metal palate. The study aimed to determine whether an acrylic palate would provide better sensory feedback and improved oral function. Participants wore each denture and completed a questionnaire. The study's results have implications for the design of complete dentures, as they highlight the importance of considering patient experiences and feedback when selecting materials. By prioritizing patient satisfaction and oral health-related quality of life, dental professionals can enhance denture treatments' effectiveness and improve patients' quality of life.

DETAILED DESCRIPTION:
Conventional dentures have long been criticized for their discomfort and limitations in oral functionality, primarily attributed to the polished surfaces covering the palate and rugae areas. To address these concerns, a rigorous randomized crossover clinical trial was meticulously conducted to compare the subjective experiences of patients wearing dentures with either an acrylic or metal palate.

The primary objective of this study was to evaluate patients' satisfaction and oral health-related quality of life while wearing dentures with different palate materials. Specifically, researchers sought to ascertain whether the use of an acrylic palate could offer superior sensory feedback and enhance overall oral function compared to traditional metal palates.

Participants enrolled in the study were required to wear both types of dentures consecutively and subsequently complete a comprehensive questionnaire designed to capture their subjective experiences and perceptions. The questionnaire encompassed various aspects, including comfort, ease of speech, ability to chew and swallow, and overall satisfaction with the dentures.

ELIGIBILITY:
Eligibility Minimum Age: 45 Years Maximum Age: 80 Years Sex: All Gender-Based Inclusion: No Accepts Healthy Volunteers: Yes (if completely edentolous)

Inclusion Criteria:

* Patients seeking a set of conventional maxillary and mandibular complete dentures at the University of Jordan Hospital, either for the first time or as a replacement for previous dentures
* Patients aged between 45 and 80 years old
* Completely edentulous for at least 3 months
* Patients who approved and consented to participation

Exclusion Criteria:

- Patients with severe underlying medical conditions, including: Neuromuscular dysfunction, Auditory problems, Mental conditions, Oral pathology, Xerostomia, Tied tongue condition

- Patients who met the inclusion criteria but failed to sign a consent form

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Patients' reported overall satisfaction with their dentures | 60 days
  Patients overall satisfaction rate using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').

SECONDARY OUTCOMES:
Patients reported oral health related quality of life | 60 days
  Patients reported oral health related quality of life using the Oral Health Impact Profile for Edentulous Patients (OHIP-EDENT) Questionnaire; The OHIP-EDENT index has 20 items and uses a 0-5 scale where 0 is never and 5 is always. The minimum overall score can be 20 and maximum 100.
Patients' reported overall satisfaction with their dentures during speaking. | 60 days
  Patients overall satisfaction rate during speaking using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').
Patients' reported overall satisfaction with their dentures during eating | 60 Days
  Patients overall satisfaction rate during eating using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').
Patients' reported overall satisfaction with their dentures during drinking | 60 Days
  Patients overall satisfaction rate during drinking using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').
Patients' reported overall satisfaction with their ability to clean their dentures | 60 Days
  Patients overall satisfaction rate with their ability to clean their dentures using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').
Patients' reported overall satisfaction with their phonetics | 60 Days
  Patients' reported overall satisfaction with their phonetics using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The study data will not be made publicly available due to ethical considerations, patient privacy concerns, and institutional policies. However, aggregate results may be published in peer-reviewed journals.